CLINICAL TRIAL: NCT02302118
Title: Survival Benefit by Esophagogastrectomy Versus Extended Gastrectomy of Patients With Carcinoma of the Esophagogastric Junction
Brief Title: Esophagogastrectomy Versus Extended Gastrectomy in AEG II
Acronym: AEG-II-EG
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: AEG-II-esophagogastrectomy
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Carcinomas of the Esophagogastric Junction
Keywords: esophageal carcinoma; kardia carcinoma
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical approach: Group A: Esophagogastrectomy Group B: Extended gastrectomy
  Interventions: Procedure: Esophagogastrectomy

INTERVENTIONS:
Procedure: Esophagogastrectomy — Esophagogastrectomy

SUMMARY:
Comparison of the oncological outcome of patients who underwent esophagogastrectomy versus extended gastrectomy due to carcinomas of the esophagogastric junction (Siewert type II)

DETAILED DESCRIPTION:
The esophagogastric junction (EGJ) is an anatomical region where different tumour entities which should be treated with different surgical approaches. Carcinomas within this area cause discordance concerning the classification due to the topographical borderland between the esophagus and the stomach. The definition, classification and staging of adenocarcinomas of the esophagogastric junction (AEG) have been inconsistent and are challenging. Siewert provided a system for classifying the tumours into three types based on topographical-anatomical criteria with direct impact on therapeutic strategies and wide acceptance in Europe. Adenocarcinomas of the esophagogastric junction type I involve the distal esophagus and mostly arise in intestinal metaplasia of Barrett's esophagus; AEG type II originates at the anatomical cardia and AEG type III are subcardial gastric carcinomas infiltrating the esophagogastric junction and distal esophagus from below. The mix of esophageal and gastric classification systems and especially, the controversy of the cell of origin of AEG type II present significant difficulties in defining this entity. The 7th edition of the American Joint Committee on Cancer/Union Internationale Contre Cancer (AJCC/UICC) classification presented a new definition of AEG in 2009. A tumour is classified as esophageal as soon as it extends into the esophagus and its epicentre is located within 5cm of the esophagogastric junction. Thus, Tumours with an epicentre in the stomach and distance greater than 5cm from the esophagogastric junction (EGJ) or those within 5cm of the EGJ but without extension into the esophagus are staged as gastric carcinoma. Most of the cardia carcinomas which originally were staged according to the gastric cancer TNM classification are now staged according the esophageal carcinoma TNM classification. Accurate preoperative staging of Siewert type II tumours is a challenge. Apparently, AEG type II show a specific biology with a high rate of lymph node metastases in comparison to distal esophageal carcinomas. The optimal surgical approach ranges from extended gastrectomy to radical esophagogastrectomy. In our opinion, an esophagogastrectomy with colonic interposition could be suggested as an appropriate approach in AEG type II. Therefore, we analyzed the oncological outcome of patients who underwent esophagogastrectomy versus extended gastrectomy due to carcinomas of the esophagogastric junction (Siewert type II).

ELIGIBILITY:
Inclusion Criteria:

* Carcinoma of the esophagogastric junction (AEG type II)
* Age of Minimum 18 years

Exclusion Criteria:

* non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carcinomas of the esophagogastric junction
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jakob R Izbicki, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg Eppendorf, Hamburg, Germany